CLINICAL TRIAL: NCT00527644
Title: Clinical Evaluation of Spring-Type Laparoscopic Clip Technology
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding to complete study
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1090979
Record Dates: First submitted 2007-09-07; First posted 2007-09-11 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: biliary leaks after laparoscopic cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spring Clips (Other): Subjects will undergo laparoscopic cholecystectomy with commercially available 5 mm spring clips utilized for the ligation of the cystic duct and artery.
  Interventions: Device: 5mm spring clip

INTERVENTIONS:
Device: 5mm spring clip — Microline Pentax 5mm Visu-Loc Clip Applier
  Other Names: Visu-Loc Clip Applier; FDA Regulation Number: 21 CFR 878.4300; FDA Regulation Name: Implantable Clip; FDA Regulatory Class: II

SUMMARY:
The Visu-Loc spring clip is being used to occlude the cystic duct at the time of laparoscopic cholecystectomy. A hepato-iminodiacetic acid (HIDA) scan will be completed on post operative day one to check for biliary leaks.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate how effective the Visu-Lock clip is at preventing leakage of bile (liquid made by liver and stored in gall bladder) after gallbladder surgery. It is not known if the Visu-Lock clip stops leaks better than other clips that have been used during gallbladder surgery.

Null hypothesis: There is no difference in subclinical or clinical leak rate between spring and crush clips used for cystic duct ligation.

Alternative hypothesis: Titanium spring clips decrease the rate of subclinical or clinical biliary leak from the cystic duct stump after laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult(18 or older)
* Diagnosis of cholelithiasis or cholecystitis
* Diagnosis of choledocholithiasis or biliary dyskinesia
* scheduled fo laparoscopic cholecystectomy
* Females: NOT pregnant

Exclusion Criteria:

* Breastfeeding
* Malignancy
* Inflammatory bowel disease (IBD)
* Ulcerative colitis (UC)
* Receiving steroids
* Severe chronic obstructive pulmonary disease (COPD) or pulmonary disorder
* History of connective tissue disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Ramshaw, MD, Principal Investigator — Chief, Division of General Surgery
Locations (1):
- University of Missouri Hospital and Clinics, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spring Clips
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Spring Clips
Number analyzed (Participants) | 14
Age, Customized [Count of Participants; unit: Participants]
  > 18 years | 14
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Unknown | 14
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: No Leak, Subclinical Leak or Clinical Bile Leak on Post-operative Hepato-iminodiacetic Acid (HIDA) Scan.
Time Frame: By post op day one HIDA scan.
Measure: Count of Participants; unit: Participants
Arm/Group | Spring Clips
Number analyzed (Participants) | 14
Participants | 14

2. Secondary Outcome: Any Other Evidence of Biliary Leak. Surgeon Assessments of Device Use: Ease of Use , Deployment and Clip Security.
Time Frame: By post op day one HIDA scan.
Population: Data not collected.
Arm/Group | Spring Clips
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Spring Clips
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

LIMITATIONS AND CAVEATS:
Study was terminated before expected enrollment was reached due to insufficient funds.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No